CLINICAL TRIAL: NCT03852992
Title: The Safety and Efficacy of Fractional Ablative 10, 600nm CO2 Laser-assisted Treatments for Male Pattern Hair Loss: a Randomized Cohort Study Comparing Stand-alone Laser Treatment, Laser Assisted Drug Delivery of Minoxidil 2% Solution , and Laser Assisted Drug Delivery of Minoxidil 2% Solution Plus Self-administration of Minoxidil 5% at Home.
Brief Title: Laser Assisted Delivery of Minoxidil in Androgenetic Alopecia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed with IRB on 10/22/22
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DERM-2018-27024
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Male Pattern Hair Loss; Androgenetic Alopecia; Male Pattern Baldness
Keywords: Male Pattern Hair Loss; Androgenetic Alopecia; Male Baldness; Bald; Baldness
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Lasers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Safety Group (Experimental): will participate in one visit, receiving laser assisted delivery of minoxidil and PK data. The safety group treatments will follow dose escalation as follows:
  * Safety Participant 1: Post-laser 5mg minoxidil (0.25ml of 20mg/ml sterile solution, applied post-laser procedure)
  * Safety Participant 2: Post-laser 10mg minoxidil (0.5ml of 20mg/ml sterile solution, applied post-laser procedure)
  * Safety Participant 3: Post-laser 20mg minoxidil (1mL of 20mg/mL sterile solution, applied post-laser procedure)
  Interventions: Device: Laser; Drug: Post-laser 5mg minoxidil; Drug: Post-laser 10mg minoxidil; Drug: Post-laser 20mg minoxidil
- Placebo (Placebo Comparator): Laser: Fractional ablative, deep mode, 5% fractional coverage
  Post-Laser Saline 0.9%: 2ml of sterile saline solution applied post-laser procedure
  Interventions: Device: Laser
- Treatment A (Experimental): Laser: Fractional ablative, deep mode, 5% fractional coverage
  Post-Laser Minoxidil 2%: 2ml of 20mg/ml sterile solution, applied post-laser procedure
  Interventions: Drug: Post-Laser Minoxidil 2%
- Treatment B (Experimental): Laser: Fractional ablative, deep mode, 5% fractional coverage
  Post-Laser Minoxidil 2%: 2ml of 20mg/ml sterile solution, applied post-laser procedure
  At-Home Minoxidil 5%: 2ml of 50mg/ml foam q24 h for duration of study
  Interventions: Drug: Post-Laser Minoxidil 2%; Drug: At-Home Minoxidil 5%

INTERVENTIONS:
Drug: Post-Laser Minoxidil 2% — 2ml of 20mg/ml sterile solution, applied post-laser procedure
  Other Names: Rogaine
  Arms: Treatment A; Treatment B
Drug: At-Home Minoxidil 5% — 2ml of 50mg/ml foam q24 h for duration of study
  Other Names: Rogaine
  Arms: Treatment B
Device: Laser — Fractional ablative, deep mode, 5% fractional coverage
  Arms: Placebo; Safety Group
Drug: Post-laser 5mg minoxidil — 0.25ml of 20mg/ml sterile solution, applied post-laser procedure
  Other Names: Rogaine
  Arms: Safety Group
Drug: Post-laser 10mg minoxidil — 0.5ml of 20mg/ml sterile solution, applied post-laser procedure
  Other Names: Rogaine
  Arms: Safety Group
Drug: Post-laser 20mg minoxidil — 1ml of 20mg/ml sterile solution, applied post-laser procedure
  Other Names: Rogaine
  Arms: Safety Group

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of fractionated ablative 10,600nm CO2 laser assisted delivery of 2% minoxidil solution in the treatment of MPHL. In this cohort study, patients will randomly be assigned stand-alone laser treatment, laser assisted drug delivery of minoxidil 2% solution, and laser assisted drug delivery of minoxidil 2% solution plus at home 5% minoxidil treatment. The primary endpoints will be to assess the change from baseline in investigator and subject Hair Growth Assessments (HGA), Hair Growth Index (HGI) and the Hair Growth Satisfaction Scale (HGSS) over 8-12 weeks in each of the three groups. The secondary endpoints will be expert assessment of hair density from baseline and evaluation of safety and adverse events, and pharmacokinetic (PK) data.

DETAILED DESCRIPTION:
Male pattern hair loss (MPHL) is a common, frustrating, and difficult to manage scalp disease with few treatment options available. Though the mechanism remains unclear, minoxidil is a well-established treatment for MPHL. With the advent of laser assisted drug delivery, the investigators seek to investigate the use of laser assisted minoxidil delivery to improve bioavailability, and subsequent hair growth for subjects MPHL. With an improved clinical outcome and increased treatment efficiency, patient quality of life would be enhanced and fewer at home topical treatments with minoxidil may be required. Additionally, this study will assist in understanding the effects of stand-alone laser therapy on hair growth and may also be used as a background or framework for a growing number of studies investigating this technology as a drug delivery system.

MPHL, also known as androgenetic alopecia, is a non-scarring alopecia resulting in gradual hair loss localized to the scalp. In men, this progressive hair loss disorder results in characteristic thinning of hair over the vertex and frontal regions.1 The Hamilton-Norwood scale categorizes this typical clinical progression.2 While the pathogenesis of MPHL is not entirely elucidated, it has been proposed to be an age and hormone dependent process with dihydrotestosterone playing a significant role.2,3 Genetic factors may also contribute to the disease.4

Topical minoxidil is an FDA approved treatment for MPHL. Minoxidil 2 and 5% solution are known to increase hair regrowth in men with androgenetic alopecia.7 While the mechanism remains unknown, it has been proposed minoxidil increases the duration of anagen and vascular supply to the follicular structure.8

Topical treatments for MPHL such as minoxidil have limited efficacy, as topical delivery of medication has low bioavailability.9 With the advent of fractionated ablative and non-ablative laser technologies, more efficient drug delivery to the level of the superficial epidermis and dermis is now possible.

The outermost layer of skin, the stratum corneum, impedes the diffusion of topical medications to follicular structures in the dermis and hypodermis. 9 Ablative fractionated laser devices create vertical channels, permitting topical medication to breach the skin's top layer, the stratum corneum, and reach deep skin layers where hair follicles reside.9

Both ablative and non-ablative fractionated laser treatments augment collagen deposition and cause growth factor mediated changes to skin ultrastructure.10 Non-ablative fractionated laser therapy in MPHL patients improves hair density with and without topical administration of growth factor.10 Our proposed study confers an additional mode of treatment beyond laser-only therapy by using an ablative fractionated laser to deliver minoxidil 2% solution percutaneously.

Herein, the investigators seek to further optimize patient treatment by investigating a combination of these treatment modalities for management of MPHL. The investigators hypothesize that fractionated ablative 10,600nm CO2 laser treatment and laser assisted drug delivery of minoxidil 2% solution will result in increased hair growth. With this improved clinical outcome and increased treatment efficiency, patient quality of life will be enhanced and fewer at home topical treatments may be required.

ELIGIBILITY:
Inclusion Criteria:

1. Males ages 21-65 years old with MPHL
2. Norwood III vertex-V. The vertex scalp must be involved
3. MPHL diagnosed by a board-certified dermatologist
4. Willing to abstain from use of over the counter products and prescription products other than those supplied in the study
5. Willing to abstain from the use of non-steroidal anti-inflammatory medications, aspirin, St. Johns Wart, and high doses of Vitamin E supplementation
6. Subjects must be capable of giving informed consent
7. Willing to adhere to protocol, including scalp examinations and photography

Exclusion Criteria:

1. Allergy or intolerance to minoxidil
2. Underlying disease that might be adversely affected by minoxidil.
3. Immunosuppressed patients (history of transplantation, cancer, chemotherapy, splenectomy, HIV)
4. Application of topical immunomodulatory or immunosuppressive agent in the preceding 6 weeks
5. Systemic administration of corticosteroid or other systemic treatment (e.g. prednisone) that has immunomodulatory or other immunosuppressive mechanism of action, in the preceding 8 weeks or planned usage at any time throughout the study
6. Clinical evidence of secondary skin infection (e.g. folliculitis)
7. Other inflammatory or infectious skin disease that might interfere with evaluations during the study
8. Investigational medications within the past 30 days
9. Severe allergies manifested by a history of anaphylaxis, or history or presence of multiple severe allergies
10. Oral retinoids within the past 6 months and topical retinoid usage within the past 4 weeks
11. Patients with history of or susceptible to keloid formation
12. Finasteride or dutasteride within the past 6 weeks
13. Spironolactone within the past 6 weeks
14. Active infection
15. Lesions in the treated area suspicious for malignancy
16. Known allergy to hair dye or hair dye components
17. Relevant history of hypotension
18. Hypertension that is untreated or uncontrolled
19. Radiation or chemotherapy to the site
20. Use of topical or oral ketoconazole in the past 6 weeks
21. Hair transplants or weaves
22. Other concomitant types of history of hair loss such as telogen effluvium
23. Medical problems including HIV, connective tissue disorder, PCOS, untreated thyroid disease
24. Psychiatric disease that that may increase risks within the trial
25. Current use of tanning beds or any active tanning
26. Use of antihypertensives or vasodilators following a first-time diagnosis of hypertension within the past 6 months
27. Planned upcoming surgeries
28. Tattoo on scalp
29. Use of oral minoxidil within the past 6 months
30. History of orthostatic hypotension
31. Adults lacking capacity to consent
32. Adults who do not speak English.
33. A medical history or clinical evidence of: acute myocardial infarction, angina, cardiac disease, cardiac tamponade, cerebrovascular disease, coronary artery disease, hypotension, orthostatic hypotension, pericardial effusion, peripheral edema, heart failure, pulmonary hypertension, renal disease, renal failure, renal impairment, pregnancy, breast-feeding, children, pheochromocytoma, skin abrasion, and geriatric.

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Hair Growth Assessment (HGA) | End of trial (8-16 weeks)
  Scale indicating graded degree of change represented as no change, worse outcome, better outcome.
Hair Growth Index (HGI) | End of trial (8-16 weeks)
  Hair growth is compared from baseline by three self-report questions on a health outcome questionnaire
Change in Hair Growth Satisfaction Scale (HGSS) | Week 0, Week 4(+4), Week 8(+4)
  Hair appearance/growth is compared from baseline by five self-report questions that rank satisfaction with hair growth on a scale from -3 (very dissatisfied) to 3 (very satisfied).
Change in Investigator Global Assessment of Photography | Week 0, end of trial (8-16 weeks)
  Scale from -3 (significant worsening) to 3 (significant improvement) assessing hair loss/growth

SECONDARY OUTCOMES:
Change in Additional Investigator Global Assessment of Photography | Week 0, end of trial (8-16 weeks)
  Scale from -3 (significant worsening) to 3 (significant improvement) assessing hair loss/growth
Change in Scalp Symptom Assessments | Week 0, Week 4(+4), Week 8(+4)
  Measure 4 criteria, erythema, scaling, pruritis, and burning/stinging, on a scale from 0 (none) to 4 (severe)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No